CLINICAL TRIAL: NCT02331134
Title: Pilot Study of Tissue and Hematopoietic/Mesenchymal Stem Cell Collection for Humanized Xenograft Studies in Melanoma and Squamous Head and Neck Cancer
Brief Title: Tissue and Hematopoietic/Mesenchymal Stem Cell for Humanized Xenograft Studies in Melanoma and Squamous Head and Neck Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Karsh Family Research Fund (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 14-0842.cc; NCI-2015-00479 (Other: CTRP)
Record Dates: First submitted 2014-12-26; First posted 2015-01-06 (Estimated); Results first posted 2023-10-31 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Malignant Melanoma; Head and Neck Cancer
Keywords: Tissue; Hematopoietic Stem Cell; Melanoma; Squamous Head and Neck Cancer
MeSH Terms: conditions — Melanoma; Head and Neck Neoplasms | interventions — Filgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Melanoma, head and neck (Other): 10 μg/kg/day of Filgrastim will be given subcutaneously for 4 days
  Interventions: Drug: Filgrastim

INTERVENTIONS:
Drug: Filgrastim — Patients will receive 10 μg/kg/day of filgrastim subcutaneously in a 4-day mobilization schedule
  Other Names: Neupogen

SUMMARY:
The overall goal of this study is to develop a pre-clinical platform of melanoma and head and neck squamous cell cancer that will allow the investigators to learn more about these diseases and discover better and more individualized treatments.

DETAILED DESCRIPTION:
The main objective of this study is to establish a humanized animal model. Investigators will consent patients who have melanoma and head and neck squamous cell cancer (HNSCC) and agree to take part in this research study. They will obtain peripheral hematopoietic stem cells (HSC), blood and tumor tissue at baseline from blood and tumor samples from these patients for use in establishing tumor explants in humanized mice. Therapy results on humanized mice will be correlated with existing or newly acquired efficacy results from those same immune-based or other therapies in patients. A secondary objective is to identify pharmacodynamic markers associated with each drug and biomarkers for evidence of efficacy or lack of thereof. Where possible, subjects receiving therapy with FDA-approved drugs of interest will be asked to provide sequential blood and tumor biopsies to study the molecular and immune events that may occur as a result of drug therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Biopsy proven incurable melanoma or incurable HNSCC amenable to have biopsy and/or surgical resection of either the primary and/or locoregional metastatic site, at the University of Colorado Hospital.
2. Age ≥ 21 years old per NCI/NIH guidelines
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0. 1, or 2
4. Adequate bone marrow, hepatic and renal function:

   * Absolute neutrophil count ≥ 1,500/µL.
   * Platelets ≥ 100,000/µL.
   * Hemoglobin ≥ 9.0 g/dL.
   * Creatinine ≤ 1.5x upper limit of normal (ULN) or calculated creatinine clearance ≥ 60 mL/min.
   * Total bilirubin ≤ 1.5x ULN.
   * Aspartate Aminotransferase (AST)/Alanine Aminotransferase ( ALT) ≤ 2x ULN.
5. Measurable disease according to Response Criteria in Solid Tumors (RECIST) version 1.1.
6. O2 saturation ≥= 93% at room air.
7. Ability to understand and willingness to sign a written informed consent document

Exclusion Criteria:

1. Contraindication (absolute or relative) to granulocyte colony-stimulating factor (G-CSF) filgrastim usage:

   * known hypersensitivity to E coli-derived proteins' filgrastim, or any other component of the product.
   * Sickle cell disorders.
   * Clinically significant and active lung hemorrhagic or inflammatory disease, including but not limited to chronic obstructive pulmonary disease (COPD), autoimmune disease, and alveolar hemorrhage; or hypoxemia of any etiology requiring oxygen.
   * Clinically significant splenomegaly or splenic metastases; history of splenic rupture, recent splenic trauma or other clinically significant splenic disease that increases the risk of splenic rupture.
2. Clinically significant and active malignancy other than incurable melanoma or head and neck squamous cell cancer.
3. Known hepatitis B or C, or HIV.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2015-05-13 (Actual); Primary Completion 2018-07-06 (Actual); Study Completion 2025-03-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Jimeno, MD, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Cancer Center, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Melanoma, Head and Neck
Started | 9
Completed | 8
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Melanoma, Head and Neck
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.1 (16.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 8
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Tissue and Hematopoietic Stem Cell Collection
Description: Tissue and hematopoietic/mesenchymal stem cell will be collected from patients with melanoma and squamous head and neck cancer. These will be used to establish humanized animal model.
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Melanoma, Head and Neck
Number analyzed (Participants) | 8
Participants | 8

ADVERSE EVENTS:
Time Frame: 42 days
Arm/Group | Melanoma, Head and Neck
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 2/8
Other Adverse Events (participants affected / at risk) | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Melanoma, Head and Neck (N=8)
Cancer Cachexia (General disorders) | 1 (1)
Left Descending Coronary Artery Stenosis (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Melanoma, Head and Neck (N=8)
Acneform rash (Skin and subcutaneous tissue disorders) | 1 (2)
Anxiety (Psychiatric disorders) | 1 (1)
Arthralgia (Immune system disorders) | 3 (3)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Atrial Flutter (Cardiac disorders) | 1 (1)
Pain (General disorders) | 3 (5)
Cachexia (General disorders) | 1 (1)
Chills (Infections and infestations) | 2 (2)
Congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dysphagia (Psychiatric disorders) | 1 (2)
Alanine aminotransferase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Fatigue (General disorders) | 3 (3)
Generalized aches (Gastrointestinal disorders) | 1 (1)
Glucosuria (Renal and urinary disorders) | 1 (1)
Headache (General disorders) | 2 (2)
Hematoma (Vascular disorders) | 1 (1)
Hot flashes (General disorders) | 1 (1)
Hyperlipidemia (Metabolism and nutrition disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 2 (2)
Lymphedema (Vascular disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Neuropathy (Nervous system disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (1)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sore throat (General disorders) | 1 (1)
Stomatitis (Infections and infestations) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2017-06-01): https://cdn.clinicaltrials.gov/large-docs/34/NCT02331134/Prot_SAP_ICF_000.pdf